CLINICAL TRIAL: NCT03738293
Title: An Observational Study to Predict Neonatal Hypoglycemia Using Antenatal Continuous Glucose Monitoring Among Late Preterm Parturients Receiving Corticosteroids
Brief Title: Continuous Glucose Monitoring of Late Preterm Birth After Corticosteroids
Status: Withdrawn | Type: Observational
Why Stopped: Study was not started at site.
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: OBX0042
Record Dates: First submitted 2018-08-14; First posted 2018-11-13 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Pregnancy Preterm; Neonatal Hypoglycemia; Prematurity
Keywords: Steroid; Corticosteroid; Betamethasone; Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women undergoing late preterm birth are at high risk of delivering a newborn with neonatal hypoglycemia. The investigators plan to monitor interstitial glucose levels prior to delivery in these women in order to develop a better understanding of the relationship between maternal hyperglycemia and neonatal hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy admitted to labor and delivery between 34w0d and 36w5d
* English speaking women
* High probability of delivery in late preterm period defined by any of the following:

  1. Membrane rupture by 2 criteria (pooling, positive nitrazine, or ferning) OR leaking amniotic fluid from the cervix
  2. Preterm labor with intact membrane, defined as at least 6 uterine contractions in 60 minutes and at least: cervical dilation greater than or equal to 3cm dilated OR 80% effaced OR planned delivery by induction of labor or cesarean in no less than 24 hrs and no more than 7 days, for any indication as deemed necessary by the provider
* Received at least one dose of corticosteroid within twelve hours of enrollment

Exclusion Criteria:

* Any prior antenatal corticosteroid course in current pregnancy
* Systemic corticosteroid administration during current pregnancy
* Fetal demise or known major fetal anomaly, including cardiac anomaly or hydrops
* Maternal contraindication to betamethasone: hypersensitivity reaction to any component of the medication, idiopathic thrombocytopenic, purpura, systemic fungal infection, or current use of amphotericin B
* Diabetes, pregestational or gestational
* Preexisting plan for intrapartum monitoring of maternal glucose levels for any reason
* Delivery expected within 12 hours of randomization, because of insufficient time for corticosteroids to confer benefit, including:

  1. Ruptured membranes with cervical dilation ≥ 3cm or with more than 6 contractions per hour unless Pitocin is deferred for at least 12 hours
  2. Chorioamnionitis
  3. Cervical dilation ≥ 8cm
  4. Evidence of non-reassuring fetal status requiring immediate delivery
* To ensure that there is an adequate proportion of women presenting at 34 to 35 weeks gestation, enrollment will be restricted so that no more than 50% of the women in the trial present at 36 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women admitted in the late preterm period who are at high risk for late preterm birth and receiving betamethasone in accordance to current American College of Obstetrician and Gynecologist guidelines are screened.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Neonatal Hypoglycemia | 48 hours
  Newborn glucose level less than 40mg/dL